CLINICAL TRIAL: NCT01720901
Title: An Open, Single-Center,Single Arm Trial to Evaluate the Efficacy and Safety of Increased Dose of Icotinib in Advanced None Small Cell Lung Cancer Patients After Routine Gefitinib Therapy
Brief Title: Increased Dose of Icotinib in Advanced None Small Cell Lung Cancer Patients After Routine Gefitinib Therapy
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Accrual limitations
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD-IC-IV41
Record Dates: First submitted 2012-10-31; First posted 2012-11-02 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Icotinib (Experimental): Icotinib will be administered 250 mg one time by month, 3 times per day.
  Interventions: Drug: Icotinib

INTERVENTIONS:
Drug: Icotinib — Icotinib will be administered 250 mg one time by month, 3 times per day.
  Other Names: Conmana; BPI-2009

SUMMARY:
To evaluate the efficacy and safety of increased dose of icotinib in advanced NSCLC patients who progressed after gefitinib therapy.

DETAILED DESCRIPTION:
This single center, single arm open label study is designed to assess the safety and efficacy of using high dose of Icotinib (Conmana) as a way to treat patients with non-small cell lung cancer that progressed after routine gefitinib therapy by progression-free survival, as well as overall survival and disease control rate. The adverse events and adverse reaction are evaluated as well.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed local advanced or metastatic stage IIIB/IV NSCLC.
* Have been treated with gefitinib and achieved completed response, partial remission, or stable disease within 3 months after first dose of gefitinib.
* At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors.
* Signed and dated informed consent before the start of specific protocol procedures.

Exclusion Criteria:

* Allergic to icotinib.
* Gefitinib excepted, experience of Anti-tumor Monoclonal Antibody or small molecular compounds therapy such as erlotinib or Cetuximab.
* Severe systemic disease out of control such as unstable or uncompensated respiratory,cardiac,liver,renal diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 4.5 months
  Progression-free survival is defined as a duration from the date that first dose is given to disease progression or death.

SECONDARY OUTCOMES:
Overall survival | 12 months
  Overall survival is a duration from the date that first dose is given to the date of death.
Tumor response | 6 weeks
  Tumor response is designed by imaging according to Response Evaluation Criteria in Solid Tumors, including complete response, partial remission, stable disease as well as progressed disease.
Adverse Events | 18 months
  Adverse events will be coded in term of the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events.

CONTACTS AND LOCATIONS:
Overall Officials: Hu Chengping, M.D., Principal Investigator — Xiangya Hospital, Central-South Univercity
Locations (1):
- Xiangya Hospital, Central-South Univercity, Changsha, Hunan, China